CLINICAL TRIAL: NCT04482504
Title: Balance Disorders Related to Pregnancy
Acronym: PRST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Other Study IDs: EC/099/2019/UNBRuzinov
Record Dates: First submitted 2020-07-18; First posted 2020-07-22 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Balance, Postural; Fall; Pregnancy Related
Keywords: static posturography; Fall; pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy pregnant women: 200 healthy pregnant women in 36.-38. Week of pregnancy. The investigators involve every healthy pregnant woman in 36.-38. week of pregnancy.
  Exclusion criteria:
  1. Unwilling to participate
  2. Minors (under 18 years old)
  e) Unfamiliar with slovak language f) Multiple pregnancy g) Musculoskeletal and neurological abnormalities
  Interventions: Diagnostic Test: 3 tests: Posturography, Questionnaire, vitamin D
- non-pregnant women: 30 non-pregnant healthy control women The investigators involve every healthy non-pregnant woman.
  Exclusion criteria:
  1. Unwilling to participate
  2. Minors (under 18 years old)
  e) Unfamiliar with slovak language f) Pregnancy g) Musculoskeletal and neurological abnormalities
  Interventions: Diagnostic Test: 3 tests: Posturography, Questionnaire, vitamin D

INTERVENTIONS:
Diagnostic Test: 3 tests: Posturography, Questionnaire, vitamin D — Posturography platform Kistler 9281B Questionnaire focused on exercise activities and self-evaluation of postural stability The investigators also determine level of vitamin D in the blood.

SUMMARY:
Primary aim of this study is to evaluate postural equilibrium and risk of falls during pregnancy by comparing static postural stability between pregnant and non-pregnant control women. Secondary aim is to find out predisposing factors of falling during pregnancy using by validated questionnaires focused on exercise activities and self-evaluation of postural stability. The investigators also determine level of vitamin D in the blood.

DETAILED DESCRIPTION:
Several hormonal, anatomical and physiological changes occur in the female body during pregnancy. These changes caused by pregnancy include significant weight gain, increased ligamentous laxity and spinal lordosis, decreased neuromuscular control and abdominal muscle strength, altered biomechanics and an anterior shift in the location of the centre of mass. These alteration of pregnant woman body can lead to balance problems.

Falls during pregnancy are very common. Pregnant women especially in advanced stage of pregnancy are at higher risk of falling compared to non-pregnant women. Falls during pregnancy may cause maternal injuries such as bone fractures, joint sprains, muscle strains, head injury, rupture of internal organs, abruptio placentae, rupture of the uterus and membranes and occasionally maternal death or intrauterine fetal demise. Pregnant women are hospitalized due to a fall 2,3 times more than non-pregnant reproductive-aged women.

There is few evidence in a literature about postural stability but not about risk factors, that caused stability disorders. By determination of risk factors, the investigators can reduce number of falls in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* The investigators involve every pregnant woman in 36.-38. week of pregnancy that attending an outpatient clinic at 2nd Department of Obstetrics and Gynecology, University Hospital Bratislava and Comenius University, Bratislava, Slovak Republic.

Exclusion Criteria:

* Unwilling to participate
* Minors (under 18 years old)
* Musculoskeletal and neurological abnormalities
* Unfamiliar with slovak language
* Multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregrancy
Study Population: pregnant and non-pregnant women
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
To determine differences of postural stability between pregnant and non-pregnant women. | 1 hour
  To determine differences of postural stability between pregnant and non-pregnant women.

SECONDARY OUTCOMES:
find out predisposing factors of falling during pregnancy | 1 hour
  Secondary aim is to find out predisposing factors of falling during pregnancy using by validated questionnaires focused on exercise activities and self-evaluation of postural stability.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Obstetrics and Gynecology, University Hospital Bratislava and Comenius University, Bratislava, Slovak Republic, Bratislava, Slovensko, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided
Not yet setup.